CLINICAL TRIAL: NCT07304401
Title: Assessment of Effectiveness of Closed-loop Spinal Cord Stimulation (CL-SCS) Therapy on Pain Reduction and Improvement of Quality of Life in Patients With Chemotherapy Induced Peripheral Neuropathy
Brief Title: Evaluation of Effectiveness of Closed-loop Spinal Cord Stimulation (CL-SCS) Therapy for Treatment of Chemotherapy Induced Peripheral Neuropathy
Acronym: CIPRESS
Status: Recruiting | Type: Observational
Sponsor: Rijnstate Hospital (Other)
Collaborators: Saluda Medical Pty Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: 2025-2667
Record Dates: First submitted 2025-12-11; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Chemotherapy Induced Peripheral Neuropathy (CIPN); Neuropathic Pain
Keywords: CIPN; Chemotherapy induced peripheral neuropathy; Spinal Cord Stimulation; SCS; Closed-Loop; neuropathic pain
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with painful chemotherapy induced peripheral neuropathy (CIPN): Subjects diagnosed with painful CIPN and eligible for SCS implantation

SUMMARY:
The goal of this observational study is to learn about the effectiveness of closed-loop spinal cord stimulation (CL-SCS) therapy for treatment of painful chemotherapy induced peripheral neuropathy.

The closed-loop SCS (CL-SCS) system stimulates the nerves in the spinal cord, measures their responses and automatically adjust the stimulation level accordingly in real time for each delivered pulse.

DETAILED DESCRIPTION:
Chemotherapy induced peripheral neuropathy (CIPN) is a serious condition that is diagnosed in up to 40% of patients who require chemotherapy. Conventional treatments for painful CIPN include both pharmacological and non-pharmacological interventions, although the underlying evidence is scarce. Spinal cord stimulation is an established treatment for pain associated with painful peripheral neuropathies. Several studies demonstrate pain relief by open-loop spinal cord stimulation (SCS) in patients with painful CIPN, with a positive effect of SCS on pain and quality of life. In the Netherlands, CIPN is an accepted indication for SCS treatment and thus SCS is a regular treatment for patients with painful and refractory CIPN. The closed-loop SCS (CL-SCS) system stimulates the dorsal column in the spinal cord, measures the response through evoked compound action potentials (ECAPs), and automatically adjust the stimulation level accordingly in real time for each delivered pulse.

The current study aims to evaluate the effectiveness of closed-loop spinal cord stimulation (CL-SCS) therapy in patients with CIPN.

ELIGIBILITY:
* Subject is deemed a suitable candidate for SCS implantation and has been routinely scheduled to undergo an SCS implantation with the Evoke SCS System.
* Subject has a minimum of leg or arm pain intensity of 5/10 on the numeric rating scale (NRS) at baseline due to CIPN.
* Patients with CIPN following chemotherapy and at least 6 months post-treatment
* CIPN symptoms for a minimum duration of 3 months.
* Patient deemed to be in remission per discretion of treating oncologist
* No existing contraindications for SCS
* Subject is ≥ 18 years old.
* Subject is not pregnant or nursing.
* Subject is willing and capable of giving informed consent.
* No satisfactory treatment effect with anti-neuropathic medication or intolerable side-effects
* No satisfactory treatment effect with minimal invasive pain treatments (including ketamine or lidocaine infusion therapy)

Exclusion Criteria:

* Patient refusal to be included in study
* Patients unwilling or mentally incapable to complete the study questionnaires
* Other causes of neuropathy (for example diabetic- or small fiber neuropathy)
* Previous treatment with SCS for CIPN
* Presence of another pain syndrome unrelated to CIPN
* History of lower limb amputation or ulceration
* Body mass index (BMI) ≥ 40
* Severe psychiatric or neurological disorders
* Any other contra indication for locoregional anaesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with painful chemotherapy induced peripheral neuropathy resistent to conventional medical management. Patients are eligible for SCS implantation and are scheduled to undergo closed-loop SCS implantation.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Overall pain intensity | The difference between baseline and the evaluation at 1, 3, 6 and 12 months after SCS implantation.
  The primary effectiveness outcome measure is pain intensity measured with the Numeric Rating Scale (NRS; 0 no pain, 10 worst imaginable pain) at 1, 3, 6 and 12 months after SCS implantation.

SECONDARY OUTCOMES:
Pain intensity for the extremities (arms and/or legs) | The difference between baseline and the evaluation at 1, 3, 6 and 12 months after SCS implantation.
  Pain intensity for the arms and/or legs measured with the Numeric Rating Scale (NRS; 0 no pain, 10 worst imaginable pain).
9-Item Patient-Reported Outcomes Measurement Information System (PROMIS-29) | The difference between baseline and the evaluation 1, 3, 6 and 12 months after SCS implantation.
  Assessment of quality of life in seven health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance) all assessed using the PROMIS-29 questionnaire. PROMIS-29 is scored on a T-score metric with a mean of 50 and a standard deviation of 10 in the U.S. general population, with a higher score representing more symptoms.
CIPN-related symptoms | The change between baseline and the evaluation 1, 3, 6 and 12 months after SCS implantation.
  Assessment of CIPN-related symptoms using the European Organization for Research and Treatment of Cancer Quality of Life-Chemotherapy-Induced Peripheral Neuropathy Questionnaire (EORTC QLQ-CIPN20).
  EORTC QLQ-CIPN20 contains 20 items scored on a 4-point Likert scale for sensory, motor and autonomic symptoms. Scale scores are linearly converted to a 0-100 scale, with higher scores indicating increased symptoms.
Medication use | The change between baseline and the evaluation 1, 3, 6 and 12 months after treatment with closed-loop SCS
  Assessment of pain medication use
Patient Global Impression of Change (PGIC) | The change between baseline and the evaluation 1, 3, 6 and 12 months after SCS implantation.
  Assessment of the patient impression of global improvement with treatment using a 7-point rating scale, ranging from 1 to 7. Higher scores indicate a patient perspective of a worsening of the health condition.
Stimulation coverage and patient stimulation awareness and satisfaction | Evaluation at 1, 3, 6 and 12 months after SCS implantation
  Assessment of the percentage of stimulation coverage of the painful area, and of stimulation sensation (awareness and quality) during closed-loop spinal cord stimulator (CL-SCS) therapy
SCS stimulation pulse width | Evaluation at 1, 3, 6 and 12 months after SCS implantation.
  The pulse width in milliseconds of the active SCS stimulation program will be collected.
SCS stimulation frequency | Evaluation at 1, 3, 6 and 12 months after SCS implantation.
  Frequency of the active SCS stimulation program measured in Hertz will be collected
(Serious) adverse events | Evaluation at 1, 3, 6 and 12 months after SCS implantation
  Assessment of treatment-related complications

CONTACTS AND LOCATIONS:
Locations (5):
- Netherlands (5):
  - Rijnstate Hospital, Arnhem
  - Sint Antonius Ziekenhuis, Nieuwegein
  - Bravis Hospital, Roosendaal
  - ETZ, Tilburg
  - ASZ, Zwijndrecht

IPD SHARING:
Plan to Share IPD: No